CLINICAL TRIAL: NCT03271294
Title: Prospective Performance Analysis of the Exair(TM) Prolapse Repair System in the Treatment of Pelvic Organ Prolapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan Institution of Women's Health PC (Other)
Collaborators: Coloplast A/S (Industry)
Responsible Party: Principal Investigator, Salil Khandwala MD, Director of Urogynecology, Michigan Institution of Women's Health PC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20160000
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2017-09-05 (Actual); Status verified 2017-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic organ prolapse; Exair; Transvaginal mesh
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Exair transvaginal mesh surgery (Other): This is a prospective study done in 80 consecutive subjects who underwent the Exair transvaginal mesh surgery from June 2013 to August 2015. The subjects were followed at 4 weeks, 6 months and 12 months post-operatively. All eligible subjects underwent a detailed urogynecologic history and examination including a Pelvic Organ Prolapse Quantification system assessment (POP-Q).
  Interventions: Device: Exair Transvaginal Mesh

INTERVENTIONS:
Device: Exair Transvaginal Mesh — Exair transvaginal mesh system for the treatment of pelvic organ prolapse

SUMMARY:
The aim of the study was to assess the role of the Exair transvaginal mesh system to correct pelvic organ prolapse from a subjective and objective standpoint. Subjects treated with the Exair transvaginal mesh for prolapse between June 2013 and August 2015 was analyzed. Subjects with uterine prolapse underwent vaginal mesh hysteropexy. There were no hysterectomies done for uterine prolapse in this study. A composite score that included subjective criteria of absence of a bothersome bulge, no prolapse below the hymen and no retreatment was used to assess success.Transvaginal Exair mesh hysteropexy offers a good option for the management of large uterine prolapses precluding the need for a hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* subjects desiring surgery for stage II or greater prolapse on the Pelvic Organ Prolapse Quantification System Assessment (POP-Q) and symptoms specific to pelvic organ prolapse mainly bothersome perception of a vaginal bulge

Exclusion Criteria:

* any physical or mental limitation that precluded their participation or inability to give informed consent

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 80 (Actual)
Dates: Start 2013-04-19 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Exair transvaginal mesh procedure success in anatomy and function at 1 year | 1 year
  Subjects who underwent the Exair transvaginal mesh surgery were followed post-operatively to determine mesh procedure success at 12 months. A composite score that included subjective criteria of absence of a bothersome bulge, no prolapse below the hymen and no retreatment was used to assess success. Subjects treated with the Exair transvaginal mesh for prolapse between June 2013 and August 2015 was analyzed. The aim of the study was to assess the role of the Exair transvaginal mesh system to correct pelvic organ prolapse from a subjective and objective standpoint.